CLINICAL TRIAL: NCT07104630
Title: Pulmonary Rehabilitation in Advanced Lung Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1525
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer Stage III; Non-small Cell Lung Cancer Stage IV; Non-small Cell Lung Cancer; Lung Cancer
Keywords: Pulmonary Rehabilitation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized between the PR arm and the usual care arm. Qualitative interviews will be conducted separately and include participants in the PR arm, participants who declined the randomized portion of the study, and medical care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulmonary Rehabilitation (PR) (Experimental)
  Interventions: Behavioral: Pulmonary Rehabilitation (PR)
- Usual care (Active Comparator)
  Interventions: Other: No intervention: Usual care
- Qualitative interviews (No Intervention): A subset of PR participants, a subset of participants who decline the randomized portion of the study, and a subset of medical care providers will participate in qualitative interviews to assess attitudes and barriers to PR.

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation (PR) — Participants will complete an 8-week course of PR, administered by certified respiratory therapists. For each week of the course, participants will attend two PR sessions. Each session will review topics such as physical function, nutrition, and psychosocial health. Participants will also be given an "exercise prescription" to complete throughout the 8-week course. The "exercise prescription" will include individualized cardiopulmonary activities.
  Arms: Pulmonary Rehabilitation (PR)
Other: No intervention: Usual care — Participants will receive standard-of-care, publicly available education on Nutrition and Cancer Survivors and Physical Activity and Cancer Survivors published by the American Institute for Cancer Research.
  Arms: Usual care

SUMMARY:
This study is for people who have previously been diagnosed with advanced stage non-small cell lung cancer (NSCLC). Many people with advanced stage NSCLC have trouble breathing and feel tired. People may be eligible for this study if they have advanced stage NSCLC and feel short of breath some of the time. NSCLC survivors may also experience things like fatigue and a lower quality of life. Pulmonary rehabilitation is a type of supportive treatment that may improve these symptoms.

This study has two parts. The first part is a randomized trial where half of the participants receive eight weeks of pulmonary rehabilitation. The other half of participants do not do pulmonary rehabilitation and instead receive the treatment that their doctors would normally recommend. The purpose of this part of the research study is to understand if pulmonary rehabilitation can help people with advanced stage NSCLC have better functioning and less shortness of breath.

The other part of the research study is an interview study. The purpose of doing interviews is to understand any challenges or obstacles that people with advanced stage NSCLC may have regarding pulmonary rehabilitation, as well as oncology care providers have with their participants going to pulmonary rehabilitation.

DETAILED DESCRIPTION:
Lung cancer (LC) is the second most common cancer in the world, (1) and the third most common cancer in the United States of America (USA) (2). Because more lung cancer screenings are being done (3-5) and because there have been advances in treatments, people will all stages of LC are living longer, including those with advanced LC. Research has shown that fatigue and breathing issues are commonly experienced by LCS (6). These symptoms can hurt the long-term health and quality of life of LCS (6-8). Currently, there are not many interventions that are used to help these symptoms for LCS.

For people with non-cancer-related respiratory disease, like chronic obstructive pulmonary disease (COPD), a type of supportive treatment called pulmonary rehabilitation (PR) can improve symptoms like difficulty breathing, fatigue, difficulty exercising, and health-related quality of life (9-11). PR is a holistic treatment plan that includes a full assessment and is then personalized to fit each person's needs. This could include things like exercise training, education, and behavior change (12). PR is considered standard-of-care for people with COPD (13). PR includes physical activity, which is something that is encouraged in all cancer survivors.

There is not much research that talks about the barriers to physical activity in survivors of lung cancer, although fatigue may be one of the most significant ones (14). Doctors may also not feel comfortable encouraging physical activities in people with lung cancer due to concerns about the safety and feasibility in exercise in people with lung cancer (15). However, PR is safe and effective in people with chronic pulmonary conditions, with well-established pathways and programs for these people.

As stated above, LCS have persistent fatigue and difficulty breathing, which is often worse in people who have metastatic LC. There is limited, high-quality evidence supporting interventions designed specifically for LCS with advanced disease. PR is potentially a safe and available intervention to improve functional status in LCS with early stage disease, and more research is needed to understand its impact on LCS with metastatic NSCLC treated with modern therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed NSCLC, Stages III or IV treated with palliative intent
* Adults ≥ 18 years of age
* ECOG performance status ≤ 3
* Clinical stability: defined as no clinical/radiographic progression within the last three months
* Self-reported dyspnea, defined as score ≥ 2 on the modified Medical Research Council (mMRC) Dyspnea Scale
* Participants must be fluent in written and spoken English

Exclusion Criteria:

* Participants being treated with curative intent for locally advanced NSCLC or oligometastatic NSCLC with concurrent chemotherapy and radiation will be excluded
* Participants have evidence of clinical and/or radiographic progression
* Mental impairment leading to inability to complete study requirements
* High risk of fracture or spine instability (Mirels score ≥7 or SINS ≥7)
* Any of the following cardiac exclusion criteria:

  * Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty or stenting within the past 6 months prior to the start of radiation therapy
  * Uncontrolled arrhythmias; individuals with rate-controlled atrial fibrillation for > 1 month prior to start of radiation therapy may be eligible
  * Syncope
  * Acute myocarditis, pericarditis, or endocarditis
  * Acute pulmonary embolus or pulmonary infarction within the last 3 months
  * Acute thrombosis of lower extremities within the last 3 months
  * Suspected dissecting aneurysm
  * Pulmonary edema
  * Respiratory failure
  * Acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in functional capacity of LCS with advanced NSCLC, as measured by the 6-minute walk test (6MWT) | Baseline, 8 weeks
  The 6MWT measures the distance (in meters) that a person can walk in 6 minutes, with higher values indicating greater functional capacity
Change in self-reported dyspnea and quality of life (QoL) in LCS with advanced NSCLC, as measured by the modified Borg scale (MBS) | Baseline, 8 weeks
  The MBS is a 1-question scale that is asked after the 6MWT, where participants rank their dyspnea (difficulty breathing) on a scale of 1-10, with greater values indicating greater difficulty.
Change in self-reported dyspnea and quality of life (QoL) in LCS with advanced NSCLC, as measured by the EORTC QLQ-C30 | Baseline, 8 weeks
  The EORTC QLQ-C30 is a 30-question questionnaire that captures functional, symptom, global health status, and QoL domains. Questions are answered on a Likert scale with four choices ranging from "Not at all" to "Very much." Greater scores indicate lower quality of life.
Change in self-reported dyspnea and quality of life (QoL) in LCS with advanced NSCLC, as measured by the EORTC QLQ-LC29 | Baseline, 8 weeks
  The EORTC QLQ-LC29 is a 29-question questionnaire that captures lung cancer-related symptoms and treatment side effects. Questions are answered on a Likert scale with four choices ranging from "Not at all" to "Very much." Greater scores indicate greater symptoms and side effects.
Change in quantity of cancer-related adverse events (AEs), as measured by the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). | Baseline, 8 weeks

SECONDARY OUTCOMES:
Participants' barriers to pulmonary rehabilitation in LCS with advanced NSCLC, as measured by thematic findings from qualitative interviews | One-time interview between month 6 and 30
  Semi-structured, qualitative interviews will be completed and assessed for qualitative, thematic findings.
Thoracic oncology providers' barriers to referral to pulmonary rehabilitation, as measured by thematic findings from qualitative interviews | One-time interview between month 6 and 30
  Semi-structured, qualitative interviews will be completed and assessed for qualitative, thematic findings.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Hsu, MD, MS, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data included in the peer reviewed publication will be publicly available. No raw data will be shared.
Time Frame: At time of publication of primary endpoints or 2 years post-trial completion, whichever is sooner.
Access Criteria: Peer reviewed publication will be publicly available.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] National Lung Screening Trial Research Team. Lung Cancer Incidence and Mortality with Extended Follow-up in the National Lung Screening Trial. J Thorac Oncol. 2019 Oct;14(10):1732-1742. doi: 10.1016/j.jtho.2019.05.044. Epub 2019 Jun 28. PMID 31260833
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] Pastorino U, Silva M, Sestini S, Sabia F, Boeri M, Cantarutti A, Sverzellati N, Sozzi G, Corrao G, Marchiano A. Prolonged lung cancer screening reduced 10-year mortality in the MILD trial: new confirmation of lung cancer screening efficacy. Ann Oncol. 2019 Jul 1;30(7):1162-1169. doi: 10.1093/annonc/mdz117. PMID 30937431
- [Background] Hsu ML, Guo MZ, Olson S, Eaton C, Boulanger M, Turner M, Miller ME, Nguyen A, Szczepanek K, Shenolikar R, Feliciano JL. Lung Cancer Survivorship: Physical, Social, Emotional, and Medical Needs of NSCLC Survivors. J Natl Compr Canc Netw. 2024 Jan 4;22(1D):e237072. doi: 10.6004/jnccn.2023.7072. PMID 38176099
- [Background] Jung JY, Lee JM, Kim MS, Shim YM, Zo JI, Yun YH. Comparison of fatigue, depression, and anxiety as factors affecting posttreatment health-related quality of life in lung cancer survivors. Psychooncology. 2018 Feb;27(2):465-470. doi: 10.1002/pon.4513. Epub 2017 Aug 17. PMID 28755492
- [Background] Hsu ML, Boulanger MC, Olson S, Eaton C, Prichett L, Guo M, Miller M, Brahmer J, Forde PM, Marrone KA, Turner M, Feliciano JL. Unmet Needs, Quality of Life, and Financial Toxicity Among Survivors of Lung Cancer. JAMA Netw Open. 2024 Apr 1;7(4):e246872. doi: 10.1001/jamanetworkopen.2024.6872. PMID 38630475
- [Background] Souto-Miranda S, Rodrigues G, Spruit MA, Marques A. Pulmonary rehabilitation outcomes in individuals with chronic obstructive pulmonary disease: A systematic review. Ann Phys Rehabil Med. 2022 May;65(3):101564. doi: 10.1016/j.rehab.2021.101564. Epub 2021 Nov 15. PMID 34329794
- [Background] Zhang H, Hu D, Xu Y, Wu L, Lou L. Effect of pulmonary rehabilitation in patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis of randomized controlled trials. Ann Med. 2022 Dec;54(1):262-273. doi: 10.1080/07853890.2021.1999494. PMID 35037535
- [Background] Troosters T, Casaburi R, Gosselink R, Decramer M. Pulmonary rehabilitation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Jul 1;172(1):19-38. doi: 10.1164/rccm.200408-1109SO. Epub 2005 Mar 18. No abstract available. PMID 15778487
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Rochester CL, Alison JA, Carlin B, Jenkins AR, Cox NS, Bauldoff G, Bhatt SP, Bourbeau J, Burtin C, Camp PG, Cascino TM, Dorney Koppel GA, Garvey C, Goldstein R, Harris D, Houchen-Wolloff L, Limberg T, Lindenauer PK, Moy ML, Ryerson CJ, Singh SJ, Steiner M, Tappan RS, Yohannes AM, Holland AE. Pulmonary Rehabilitation for Adults with Chronic Respiratory Disease: An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2023 Aug 15;208(4):e7-e26. doi: 10.1164/rccm.202306-1066ST. PMID 37581410
- [Background] Ng AH, Ngo-Huang A, Vidal M, Reyes-Garcia A, Liu DD, Williams JL, Fu JB, Yadav R, Bruera E. Exercise Barriers and Adherence to Recommendations in Patients With Cancer. JCO Oncol Pract. 2021 Jul;17(7):e972-e981. doi: 10.1200/OP.20.00625. Epub 2021 Mar 19. PMID 33739853
- [Background] Granger CL, Denehy L, Remedios L, Retica S, Phongpagdi P, Hart N, Parry SM. Barriers to Translation of Physical Activity into the Lung Cancer Model of Care. A Qualitative Study of Clinicians' Perspectives. Ann Am Thorac Soc. 2016 Dec;13(12):2215-2222. doi: 10.1513/AnnalsATS.201607-540OC. PMID 27689958